CLINICAL TRIAL: NCT02476253
Title: Sodium Bicarbonate to Treat Severe Acidosis in the Critically Ill : A Multiple Center Randomized Clinical Trial (BICAR-ICU)
Brief Title: Sodium Bicarbonate to Treat Severe Acidosis in the Critically Ill
Acronym: (BICAR-ICU)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9260
Record Dates: First submitted 2015-06-10; First posted 2015-06-19 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2017-06

CONDITIONS: Metabolic Acidosis
Keywords: acidosis; shock; sodium bicarbonate; renal replacement therapy
MeSH Terms: conditions — Acidosis; Shock | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intravenous 4.2% Sodium Bicarbonate 125ml to 250ml / 30min up to 1000ml/24h to maintain plasma pH equal or greater than 7.30
  Interventions: Drug: Sodium Bicarbonate
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Sodium Bicarbonate — Intravenous 4.2% Sodium Bicarbonate 125ml to 250ml / 30min up to 1000ml/24h to maintain plasma pH equal or greater than 7.30
  Arms: Intervention

SUMMARY:
The purpose of the present study is to compare the adjunct treatment of metabolic or mixed severe acidosis in the critically ill using Sodium Bicarbonate as a buffer to increase the plasma pH vs no buffering therapy.

The study is a randomized multiple center clinical trial with the outcome as a primary endpoint.

DETAILED DESCRIPTION:
* Design: randomized multiple center clinical trial, open label
* Arms: intravenous 4.2% Sodium Bicarbonate vs no additional treatment
* Inclusion: age of 18 yo or above, critically ill patient with a SOFA score of 4 or above, lactatemia of 2mmol/l or above, with pH of 7.20 or below and PaCO2 of 45mmHg or below and bicarbonatemia of 20mmol/l or below
* Exclusion: single respiratory disorder (PaCO2 > 50 mmHg, Bicarbonatemia equal or higher than (PaCO2-40)/10 + 24 ; acute diarrhea, ileostomy or biliary drainage ; stage IV kidney failure or chronic dialysis ; tubular acidosis, ketoacidosis, high anion gap acids poisoning (PEG, aspirin, methanol) ; PaCO2 equal to 45mmHg or above and spontaneous breathing, pregnancy, protected patients, moribund patient (life expectancy of 48h or below)
* Randomization: website randomization with stratification on age, presence of sepsis at inclusion, renal failure
* Intervention: experimental arm: intravenous 4.2% Sodium Bicarbonate 125 to 250ml in 30min up to 1000ml/24h. The target is a plasma pH of 7.30 or above.
* An interim statistical analysis is planned when 200 patients will be included

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 yo or above,
* Critically ill patient with a SOFA score of 4 or above,
* Lactatemia of 2mmol/l or above, with pH of 7.20 or below and PaCO2 of 45mmHg or below and bicarbonatemia of 20mmol/l or below

Exclusion Criteria:

* Administration of Sodium Bicarbonate 24 hours before inclusion
* Single respiratory disorder (PaCO2 > 50 mmHg, Bicarbonatemia equal or higher than (PaCO2-40)/10 + 24
* Acute diarrhea, ileostomy or biliary drainage
* Stage IV kidney failure or chronic dialysis
* Tubular acidosis, ketoacidosis, high anion gap acids poisoning (PEG, aspirin, methanol)
* PaCO2 equal to 45mmHg or above and spontaneous breathing, pregnancy, protected patients, moribund patient (life expectancy of 48h or below)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Composite criteria of Day 28 mortality and/or patients with at least one organ failure defined as a SOFA score of 3 or 4 | Day 0 to Day 28
  Composite criteria of Day 28 mortality and/or patients with at least one organ failure defined as a SOFA score of 3 or 4

SECONDARY OUTCOMES:
Evolution of the organ failure scores | Day 0 to Day 28
  use of SOFA score to assess the outcome 2
Duration of renal replacement therapy (days) | Day 0 to Day 28
  need to renal replacement therapy
Duration of mechanical ventilation and ventilatory free days (days) | Day 0 to Day 28
  duration of mechanical ventilation and ventilatory free days
Duration of vasopressors administration (h) | Day 0 to Day 28
  need for vasopressors and fluids using duration of vasopressor infusion (D0 to D28)
Hospital acquired infections (incidence) | Day 0 to Day 28
  hospital acquired infections using United States Centers for Disease Control definitions and a dedicated document
Amount of intravenous fluid (ml) | Day 0 to Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- DAR St Eloi, Montpellier, France

REFERENCES:
- [Background] Kellum JA, Levin N, Bouman C, Lameire N. Developing a consensus classification system for acute renal failure. Curr Opin Crit Care. 2002 Dec;8(6):509-14. doi: 10.1097/00075198-200212000-00005. PMID 12454534
- [Background] Dubin A, Menises MM, Masevicius FD, Moseinco MC, Kutscherauer DO, Ventrice E, Laffaire E, Estenssoro E. Comparison of three different methods of evaluation of metabolic acid-base disorders. Crit Care Med. 2007 May;35(5):1264-70. doi: 10.1097/01.CCM.0000259536.11943.90. PMID 17334252
- [Background] Smith I, Kumar P, Molloy S, Rhodes A, Newman PJ, Grounds RM, Bennett ED. Base excess and lactate as prognostic indicators for patients admitted to intensive care. Intensive Care Med. 2001 Jan;27(1):74-83. doi: 10.1007/s001340051352. PMID 11280677
- [Background] Gunnerson KJ, Saul M, He S, Kellum JA. Lactate versus non-lactate metabolic acidosis: a retrospective outcome evaluation of critically ill patients. Crit Care. 2006 Feb;10(1):R22. doi: 10.1186/cc3987. PMID 16507145
- [Background] Jung B, Rimmele T, Le Goff C, Chanques G, Corne P, Jonquet O, Muller L, Lefrant JY, Guervilly C, Papazian L, Allaouchiche B, Jaber S; AzuRea Group. Severe metabolic or mixed acidemia on intensive care unit admission: incidence, prognosis and administration of buffer therapy. A prospective, multiple-center study. Crit Care. 2011;15(5):R238. doi: 10.1186/cc10487. Epub 2011 Oct 13. PMID 21995879
- [Background] Husain FA, Martin MJ, Mullenix PS, Steele SR, Elliott DC. Serum lactate and base deficit as predictors of mortality and morbidity. Am J Surg. 2003 May;185(5):485-91. doi: 10.1016/s0002-9610(03)00044-8. PMID 12727572
- [Background] Kellum JA. Clinical review: reunification of acid-base physiology. Crit Care. 2005 Oct 5;9(5):500-7. doi: 10.1186/cc3789. Epub 2005 Aug 5. PMID 16277739
- [Background] Forsythe SM, Schmidt GA. Sodium bicarbonate for the treatment of lactic acidosis. Chest. 2000 Jan;117(1):260-7. doi: 10.1378/chest.117.1.260. PMID 10631227
- [Background] Fencl V, Jabor A, Kazda A, Figge J. Diagnosis of metabolic acid-base disturbances in critically ill patients. Am J Respir Crit Care Med. 2000 Dec;162(6):2246-51. doi: 10.1164/ajrccm.162.6.9904099. PMID 11112147
- [Background] Kellum JA, Song M, Almasri E. Hyperchloremic acidosis increases circulating inflammatory molecules in experimental sepsis. Chest. 2006 Oct;130(4):962-7. doi: 10.1378/chest.130.4.962. PMID 17035425
- [Background] Kellum JA, Song M, Venkataraman R. Effects of hyperchloremic acidosis on arterial pressure and circulating inflammatory molecules in experimental sepsis. Chest. 2004 Jan;125(1):243-8. doi: 10.1378/chest.125.1.243. PMID 14718447
- [Background] Morimoto Y, Morimoto Y, Kemmotsu O, Alojado ES. Extracellular acidosis delays cell death against glucose-oxygen deprivation in neuroblastoma x glioma hybrid cells. Crit Care Med. 1997 May;25(5):841-7. doi: 10.1097/00003246-199705000-00021. PMID 9187605
- [Background] Laffey JG, O'Croinin D, McLoughlin P, Kavanagh BP. Permissive hypercapnia--role in protective lung ventilatory strategies. Intensive Care Med. 2004 Mar;30(3):347-56. doi: 10.1007/s00134-003-2051-1. Epub 2004 Jan 14. PMID 14722644
- [Background] Kraut JA, Madias NE. Metabolic acidosis: pathophysiology, diagnosis and management. Nat Rev Nephrol. 2010 May;6(5):274-85. doi: 10.1038/nrneph.2010.33. Epub 2010 Mar 23. PMID 20308999
- [Background] Cohen MV, Yang XM, Downey JM. The pH hypothesis of postconditioning: staccato reperfusion reintroduces oxygen and perpetuates myocardial acidosis. Circulation. 2007 Apr 10;115(14):1895-903. doi: 10.1161/CIRCULATIONAHA.106.675710. Epub 2007 Mar 26. PMID 17389262
- [Background] Bersin RM, Chatterjee K, Arieff AI. Metabolic and hemodynamic consequences of sodium bicarbonate administration in patients with heart disease. Am J Med. 1989 Jul;87(1):7-14. doi: 10.1016/s0002-9343(89)80476-0. PMID 2741982
- [Background] Cooper DJ, Walley KR, Wiggs BR, Russell JA. Bicarbonate does not improve hemodynamics in critically ill patients who have lactic acidosis. A prospective, controlled clinical study. Ann Intern Med. 1990 Apr 1;112(7):492-8. doi: 10.7326/0003-4819-112-7-492. PMID 2156475
- [Background] Mathieu D, Neviere R, Billard V, Fleyfel M, Wattel F. Effects of bicarbonate therapy on hemodynamics and tissue oxygenation in patients with lactic acidosis: a prospective, controlled clinical study. Crit Care Med. 1991 Nov;19(11):1352-6. doi: 10.1097/00003246-199111000-00008. PMID 1935152
- [Background] El-Solh AA, Abou Jaoude P, Porhomayon J. Bicarbonate therapy in the treatment of septic shock: a second look. Intern Emerg Med. 2010 Aug;5(4):341-7. doi: 10.1007/s11739-010-0351-3. Epub 2010 Feb 19. PMID 20169423
- [Background] Fang ZX, Li YF, Zhou XQ, Zhang Z, Zhang JS, Xia HM, Xing GP, Shu WP, Shen L, Yin GQ. Effects of resuscitation with crystalloid fluids on cardiac function in patients with severe sepsis. BMC Infect Dis. 2008 Apr 17;8:50. doi: 10.1186/1471-2334-8-50. PMID 18419825
- [Background] Kraut JA, Kurtz I. Use of base in the treatment of acute severe organic acidosis by nephrologists and critical care physicians: results of an online survey. Clin Exp Nephrol. 2006 Jun;10(2):111-7. doi: 10.1007/s10157-006-0408-9. PMID 16791396
- [Background] Kellum JA. Disorders of acid-base balance. Crit Care Med. 2007 Nov;35(11):2630-6. doi: 10.1097/01.CCM.0000286399.21008.64. PMID 17893626
- [Background] Kraut JA, Kurtz I. Metabolic acidosis of CKD: diagnosis, clinical characteristics, and treatment. Am J Kidney Dis. 2005 Jun;45(6):978-93. doi: 10.1053/j.ajkd.2005.03.003. PMID 15957126
- [Background] Shah SN, Abramowitz M, Hostetter TH, Melamed ML. Serum bicarbonate levels and the progression of kidney disease: a cohort study. Am J Kidney Dis. 2009 Aug;54(2):270-7. doi: 10.1053/j.ajkd.2009.02.014. Epub 2009 Apr 25. PMID 19394734
- [Background] Brar SS, Shen AY, Jorgensen MB, Kotlewski A, Aharonian VJ, Desai N, Ree M, Shah AI, Burchette RJ. Sodium bicarbonate vs sodium chloride for the prevention of contrast medium-induced nephropathy in patients undergoing coronary angiography: a randomized trial. JAMA. 2008 Sep 3;300(9):1038-46. doi: 10.1001/jama.300.9.1038. PMID 18768415
- [Background] Kelly AM, Dwamena B, Cronin P, Bernstein SJ, Carlos RC. Meta-analysis: effectiveness of drugs for preventing contrast-induced nephropathy. Ann Intern Med. 2008 Feb 19;148(4):284-94. doi: 10.7326/0003-4819-148-4-200802190-00007. PMID 18283206
- [Background] From AM, Bartholmai BJ, Williams AW, Cha SS, Pflueger A, McDonald FS. Sodium bicarbonate is associated with an increased incidence of contrast nephropathy: a retrospective cohort study of 7977 patients at mayo clinic. Clin J Am Soc Nephrol. 2008 Jan;3(1):10-8. doi: 10.2215/CJN.03100707. Epub 2007 Dec 5. PMID 18057306
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Background] Brochard L, Abroug F, Brenner M, Broccard AF, Danner RL, Ferrer M, Laghi F, Magder S, Papazian L, Pelosi P, Polderman KH; ATS/ERS/ESICM/SCCM/SRLF Ad Hoc Committee on Acute Renal Failure. An Official ATS/ERS/ESICM/SCCM/SRLF Statement: Prevention and Management of Acute Renal Failure in the ICU Patient: an international consensus conference in intensive care medicine. Am J Respir Crit Care Med. 2010 May 15;181(10):1128-55. doi: 10.1164/rccm.200711-1664ST. PMID 20460549
- [Background] Ferrer M, Sellares J, Valencia M, Carrillo A, Gonzalez G, Badia JR, Nicolas JM, Torres A. Non-invasive ventilation after extubation in hypercapnic patients with chronic respiratory disorders: randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1082-8. doi: 10.1016/S0140-6736(09)61038-2. Epub 2009 Aug 12. PMID 19682735
- [Background] RENAL Replacement Therapy Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lo S, McArthur C, McGuinness S, Myburgh J, Norton R, Scheinkestel C, Su S. Intensity of continuous renal-replacement therapy in critically ill patients. N Engl J Med. 2009 Oct 22;361(17):1627-38. doi: 10.1056/NEJMoa0902413. PMID 19846848
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Jaber S, Jung B, Sebbane M, Ramonatxo M, Capdevila X, Mercier J, Eledjam JJ, Matecki S. Alteration of the piglet diaphragm contractility in vivo and its recovery after acute hypercapnia. Anesthesiology. 2008 Apr;108(4):651-8. doi: 10.1097/ALN.0b013e31816725a6. PMID 18362597
- [Background] Ichai C, Massa H, Hubert S. c. In: SAS EM, editor. EMC Anesthésie-Réanimation. Paris; 2006.
- [Background] Correction de l'acidose métabolique en réanimation. 1999 [cited; Available from: http://www.urgences-serveur.fr/IMG/pdf/correction_acidose.pdf
- [Derived] Jaber S, Paugam C, Futier E, Lefrant JY, Lasocki S, Lescot T, Pottecher J, Demoule A, Ferrandiere M, Asehnoune K, Dellamonica J, Velly L, Abback PS, de Jong A, Brunot V, Belafia F, Roquilly A, Chanques G, Muller L, Constantin JM, Bertet H, Klouche K, Molinari N, Jung B; BICAR-ICU Study Group. Sodium bicarbonate therapy for patients with severe metabolic acidaemia in the intensive care unit (BICAR-ICU): a multicentre, open-label, randomised controlled, phase 3 trial. Lancet. 2018 Jul 7;392(10141):31-40. doi: 10.1016/S0140-6736(18)31080-8. Epub 2018 Jun 14. PMID 29910040